CLINICAL TRIAL: NCT03485950
Title: An Investigator Initiated, Phase II Single-Center, Randomized, Open-Label, Prospective, Comparative Study to Determine the Efficacy, Safety, and Tolerability of Ceftolozane-Tazobactam Plus Vancomycin, Linezolid Versus Standard of Care Plus Vancomycin, Linezolid as Empiric Therapy in Febrile Neutropenic Adults With Cancer
Brief Title: Comparative Study To Determine The Efficacy, Safety, And Tolerability Of Ceftolozane-Tazobactam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0729; NCI-2018-00755 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0729 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-03-26; First posted 2018-04-03 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Other Infectious Diseases
Keywords: Other infectious diseases; Febrile neutropenic adults with cancer; Ceftolozane-Tazobactam; Cefepime; Meropenem; Piperacillin/Tazobactam
MeSH Terms: interventions — Cefepime; ceftolozane; Meropenem; Piperacillin, Tazobactam Drug Combination; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (ceftolozane-tazobactam) (Experimental): Participants receive ceftolozane-tazobactam IV over 1 hour every 8 hours for up to 14 days in the absence of disease progression or unacceptable toxicity. After at least 3 days, participants may switch to different PO or IV antibiotics at the discretion of the study doctor.
  Interventions: Drug: Ceftolozane; Other: Laboratory Biomarker Analysis; Drug: Tazobactam
- Group II (standard of care antibiotic treatment) (Active Comparator): Participants receive standard of care antibiotic treatment consisting of either cefepime IV over 30 minutes every 8 hours, meropenem IV over 30 minutes every 8 hours, or piperacillin-tazobactam IV over 1 hour every 6 hours for up to 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cefepime; Other: Laboratory Biomarker Analysis; Drug: Meropenem; Drug: Piperacillin-Tazobactam; Drug: Tazobactam

INTERVENTIONS:
Drug: Cefepime — Given IV
  Arms: Group II (standard of care antibiotic treatment)
Drug: Ceftolozane — Given IV
  Other Names: CXA-101
  Arms: Group I (ceftolozane-tazobactam)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Meropenem — Given IV
  Other Names: Meropenem Trihydrate; Merrem I.V.; SM-7338
  Arms: Group II (standard of care antibiotic treatment)
Drug: Piperacillin-Tazobactam — Given IV
  Other Names: PIPER/TAZO; Piperacillin/Tazobactam; Zosyn
  Arms: Group II (standard of care antibiotic treatment)
Drug: Tazobactam — Given IV
  Other Names: YTR-830H

SUMMARY:
The goal of this clinical research study is to learn if the study drug ceftolozane-tazobactam is more effective in controlling febrile neutropenia (fever and low white blood cell counts) than using approved antibiotics in patients with cancer. The safety of ceftolozane-tazobactam will also be studied.

This is an investigational study. Ceftolozane-tazobactam is FDA approved and commercially available to treat certain types of infections. It is not approved for the treatment of febrile neutropenia, either by itself or in combination with other antibiotics. Its use to treat febrile neutropenia is investigational.

All other antibiotics given on this study are FDA approved and commercially available for the treatment of infections. However, only cefepime is specifically FDA approved to treat febrile neutropenia. The study doctor can explain how the study drugs are designed to work.

Up to 100 participants will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Groups and Study Drug Administration:

If participant is found to be eligible to take part in this study and participant agrees, participant will be randomly assigned (as in the flip of a coin) to either receive either the study drug (Group 1) or a standard treatment antibiotic (Group 2). This is done because no one knows if one study group is better, the same, or worse than the other group. Both participant and the study doctor will know what participant is receiving.

If participant is in Group 1, participant will receive ceftolozane-tazobactam by vein over 1 hour every 8 hours.

If participant is in Group 2, participant will receive a standard treatment antibiotic. This may include one of the following 3 options:

cefepime by vein over about 30 minutes every 8 hours. meropenem by vein over about 30 minutes every 8 hours. piperacillin/tazobactam by vein over about 1 hour every 6 hours.

Participant will receive the study drugs by vein for at least 3 days. After 3 days, if the study doctor thinks it is in participant's best interest and participant is eligible, participant may switch to receiving a different antibiotic either by mouth or by vein. The study doctor will tell participant more about what antibiotic participant may begin to receive, how it is administered, and its possible risks. If participant begins taking the study drugs by mouth, the study doctor or study staff will tell participant how and when to take each drug.

If the doctor thinks it is needed, participant will be given additional standard drugs to help control the infection. Participant may ask the study staff for information about how the drugs are given and their risks.

Length of Study:

Participant may receive the study drugs for up to 14 days. Participant will no longer be able to receive the study drugs if the disease gets worse, if intolerable side effects occur, if participant needs treatment that is not allowed on this study, or if participant is unable to follow study directions.

Participation on this study will be over after the late follow-up visit.

Study Visits:

Participant will have the following tests/procedures while participant is in the hospital. If participant begins to take the study drugs by mouth, participant will no longer have these study visits.

Each day for up to 2 weeks, if the doctor thinks it is needed, blood (about 1 tablespoon) or urine will be collected for routine tests.

Every 2 days for up to 2 weeks, blood (about 1 tablespoon) will be drawn to check for infection. Participant will stop having these blood draws when there is no longer a sign of infection and participant does not have a fever.

Twice each week for up to 2 weeks, participant will have a physical exam.

Follow-Up:

Within 72 hours (3 days) after participant's last dose of participant's assigned study treatment and before starting the second antibiotic therapy (if applicable):

Participant will have a physical exam. Blood (about 1 tablespoon) and urine will be collected for routine tests. If participant tested positive for infection at the beginning of the study, blood (about 1 tablespoon) will be drawn to check for infection. The study doctor will tell participant if participant will have this blood draw.

About 21-28 days (3-4 weeks) after participant's first dose of study drug, participant will return to MD Anderson for the following tests/procedures:

Participant will have a physical exam. If participant tested positive for infection at the beginning of the study, blood (about 1 tablespoon) will be drawn to check for infection. The study doctor will tell participant if participant will have this blood draw.

If participant can become pregnant, blood (about 1 teaspoon) will be drawn for a pregnancy test.

About 35-42 days (5-6 weeks) after participant's first dose of study drug, a member of the study staff will call participant to ask about any new drugs participant may have started and if participant is having any side effects. If participant is called, it should last about 10 minutes. If the doctor or study staff thinks it is needed, participant will be asked to come back to the clinic for the following tests/procedures:

Participant will have a physical exam. If the doctor thinks it is needed, blood (about 1 tablespoon) will be drawn to check for infection.

At any of these follow-up visits, if participant's doctor thinks it is needed, participant will have a chest x-ray or CT scan to check participant's lungs.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent, and has the willingness and ability to comply with all study procedures
* Patients with neutropenic fever who have existing malignancy or have undergone hematopoietic stem cell transplantation; neutropenic fever is defined as the presence of neutropenia defined by: 1) absolute neutrophil count (ANC) < 500 cells/mm^3 or has an ANC that is expected to decrease to < 500 cells/mm^3 within 48 hours of trial entry and fever defined as: 2) single oral temperature measurement of > 101 degree Fahrenheit (F) (38.3 degree Celsius [C]) or a temperature of > 100.4 degree F (38.0 degree C) sustained over a 1-hour period
* Requires hospitalization for IV empiric antibiotic therapy
* If female: not breastfeeding; agrees to not attempt to become pregnant during the study; is surgically sterile or at least 2-years postmenopausal, or if of childbearing potential, has negative screening serum pregnancy test (if serum pregnancy test results are not available at the time of enrollment, a negative urine pregnancy test is required within 24 hours.); if of childbearing potential (including being < 2 years postmenopausal), is willing to practice sexual abstinence or use an effective dual form of contraception with her partner (eg, 2 barrier methods, barrier method plus hormonal method) during treatment and for ≥ 28 days after the last dose of any study therapy (IV or oral)

Exclusion Criteria:

* History of any hypersensitivity or allergic reaction to any cephalosporin antibiotic or tazobactam
* Fever suspected to be caused by a noninfectious cause (eg, fever related to drug or blood product administration)
* Confirmed fungal infection (eg, Pneumocystis jirovecii etiology in patients with pneumonia) that justifies adding additional empiric antimicrobial therapy (eg, antifungals)
* Confirmed viral infection that justifies adding additional empiric antiviral therapy (eg, ganciclovir, foscarnet)
* Known acute viral hepatitis
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level > 5 times the upper limit of normal (x ULN); patients with values > 3 x ULN and < 5 x ULN are eligible if the value is acute and directly related to the infectious process being treated
* Total bilirubin > 3 x ULN unless isolated hyperbilirubinemia is directly related to the acute infection or due to known Gilbert disease; manifestations of end-stage liver disease, such as ascites or hepatic encephalopathy
* Known to be human immunodeficiency virus positive
* Severely impaired renal function, defined as creatinine clearance (CrCl) =< 30 mL/min estimated by the Cockcroft-Gault formula
* Expected requirement for hemodialysis while on study therapy
* Received > 24 hours of IV antibacterial therapy (with study drugs) within 72 hours of the initiation of inpatient IV study drug for treatment of suspected infection; antibiotic prophylaxis and oral antibiotics is allowed; prophylactic use of antiviral or antifungal medication is permitted
* Requirement for any non-study potentially effective concomitant systemic antibacterial therapy
* Past or current history of epilepsy or seizure disorder; exception: well-documented febrile seizure of childhood
* Evidence of immediately life-threatening disease, progressively fatal disease, or life expectancy of 3 months or less (eg, moribund or with shock unresponsive to fluid replacement)
* Unable or unwilling to adhere to the study-specified procedures and restrictions
* Any condition that would make the patient, in the opinion of the investigator, unsuitable for the study (eg, would place a patient at risk or compromise the quality of the data
* Participation in any other ongoing ceftolozane/tazobactam trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam I Raad, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chaftari AM, Hachem R, Malek AE, Mulanovich VE, Szvalb AD, Jiang Y, Yuan Y, Ali S, Deeba R, Chaftari P, Raad I. A Prospective Randomized Study Comparing Ceftolozane/Tazobactam to Standard of Care in the Management of Neutropenia and Fever in Patients With Hematological Malignancies. Open Forum Infect Dis. 2022 Feb 14;9(6):ofac079. doi: 10.1093/ofid/ofac079. eCollection 2022 Jun. PMID 35663286
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceftolozane/Tazobactam Arm: Received IV Ceftolozane/Tazobactam (minimum of 9 doses). Patients may receive other additional therapy.
- Standard of Care (SOC) Arm: Received one of the following IV therapies: Cefepime (minimum of 9 doses), Meropenem (minimum of 9 doses), Piperacillin/Tazobactam (minimum of 12 doses). Patients may receive other additional therapy.
Period: Overall Study
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Started | 50 | 50
Completed | 43 | 48
Not Completed | 7 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: Patients in Modified Intent-To-Treat (MITT) analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm | Total
Number analyzed (Participants) | 47 | 50 | 97
Age, Continuous [Median (Full Range); unit: years] | 60 [25 to 84] | 55 [18 to 79] | 56 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 28 | 32 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 4 | 5 | 9
  Hispanic or Latino | 6 | 7 | 13
  Middle East | 3 | 1 | 4
  White | 32 | 35 | 67
  Others | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 47 | 50 | 97
Type of Hematological malignancy [Count of Participants; unit: Participants]
  Acute Lymphocytic Leukemia(ALL) | 9 | 12 | 21
  Chronic Lymphocytic Leukemia (AML) | 19 | 22 | 41
  Chronic Myeloid Leukemia (CML) | 3 | 0 | 3
  Lymphoma | 9 | 6 | 15
  Others | 7 | 10 | 17
History of Bone Marrow Transplant (BMT) within 1 year [Count of Participants; unit: Participants]
  Autologous | 2 | 4 | 6
  Allogeneic | 4 | 5 | 9
Temperature at initial presentation [Count of Participants; unit: Participants]
  < 36 Celsius | 0 | 0 | 0
  36 -38 Celsius | 3 | 7 | 10
  >38 Celsius | 44 | 43 | 87
Site of Microorganisms [Count of Participants; unit: Participants]
  Genitourinary | 2 | 1 | 3
  Blood | 10 | 12 | 22
Organism of positive culture [Count of Participants; unit: Participants]
  Entereococcus faecalis | 0 | 2 | 2
  E. coli | 0 | 2 | 2
  Klebsiella pneumoniae | 1 | 0 | 1
  Methicillin-resistant Staphylococcus aureus (MRSA) | 2 | 1 | 3
  Pseudomonas aeruginosa | 1 | 0 | 1
  Rothia mucilaginous | 1 | 0 | 1
  Streptococcus viridans | 5 | 5 | 10
  Staphylococcus epidermidis | 0 | 2 | 2
  Entereococcus faecalis + E coli | 1 | 0 | 1
  Enterococcus faecalis + Pseudomonas aeruginosa | 1 | 0 | 1
Temperature at baseline [Median (Inter-Quartile Range); unit: Celsius] | 37.3 [36.9 to 38.2] | 37.5 [37.0 to 38.3] | 37.4 [37.0 to 38.3]
Microbiology Documentation [Count of Participants; unit: Participants] — Site of Microorganisms
  Participants
    Genitourinary | 2 | 0 | 2
    Blood | 10 | 11 | 21
    Genitourinary and Blood | 0 | 1 | 1
Bacterial Pathogen Causing Documented Infection [Count of Participants; unit: Participants]
  Gram Negative | 2 | 2 | 4
  Gram Negative and Gram Positive | 2 | 0 | 2
  Gram Positive | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Favorable Clinical Response at End of Inpatient Intravenous Therapy (EOIV)
Description: Resolution of all acute signs and symptoms of the primary infection or improvement to such an extent that no additional antibacterial therapy is required (ie, except for protocol-allowed adjunctive therapies and/or oral or IV switch) and such that no more than 14 days of total antibacterial therapy is required.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug
Population: Patients in MITT (Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 47 | 50
Participants | 41 | 36

2. Secondary Outcome: Number of Participants With Favorable Clinical Response in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set at EOIV.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at end of inpatient intravenous therapy (EOIV). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug.
Population: Patients in mMITT (Microbiological Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 4 | 2
Participants | 3 | 1

3. Secondary Outcome: Number of Participants With Favorable Clinical Response in the Clinically Evaluable (CE) Analysis Set at EOIV.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the CE (Clinically Evaluable) Analysis Set at end of inpatient intravenous therapy (EOIV). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug.
Population: Patients in CE (Clinically Evaluable) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 31 | 38
Participants | 29 | 32

4. Secondary Outcome: Number of Participants With Favorable Clinical Response in the MITT Analysis Set at TOC
Description: The secondary efficacy outcome is favorable clinical response of the patients in the MITT (Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug
Population: Patients in the MITT (Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 47 | 50
Participants | 34 | 28

5. Secondary Outcome: Number of Participants With Favorable Clinical Response in the MITT Analysis Set at Late Follow-Up (LFU)
Description: The secondary efficacy outcome is favorable clinical response of the patients in the MITT (Modified Intent-To-Treat) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug
Population: Patients in the MITT (Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 47 | 50
Participants | 33 | 26

6. Secondary Outcome: Number of Participants With Favorable Clinical Response in the mMITT Analysis Set at Test of Cure (TOC)
Description: The secondary efficacy outcome is favorable clinical response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: Patients in mMITT (Microbiological Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 4 | 2
Participants | 3 | 1

7. Secondary Outcome: Number of Participants With Favorable Clinical Response in the mMITT Analysis Set at Late Follow-Up (LFU)
Description: The secondary efficacy outcome is favorable clinical response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug
Population: Patients in mMITT (Microbiological Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 4 | 2
Participants | 3 | 1

8. Secondary Outcome: Number of Participants With Favorable Clinical Response in the CE Analysis Set at TOC
Description: The secondary efficacy outcome is favorable clinical response of the patients in the CE (Clinically Evaluable) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug
Population: Patients in CE (Clinically Evaluable) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 31 | 38
Participants | 28 | 26

9. Secondary Outcome: Number of Participants With Favorable Clinical Response in the CE Analysis Set at LFU.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the CE (Clinically Evaluable) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug
Population: Patients in CE (Clinically Evaluable) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 31 | 38
Participants | 27 | 24

10. Secondary Outcome: Number of Participants With Favorable Clinical Response in the ME Analysis Set at EOIV.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the ME (Microbiologically Evaluable) Analysis Set at end of inpatient intravenous therapy (EOIV). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug.
Population: Patients in CE analysis set with baseline Gram-negative pathogen (= ME (Microbiologically Evaluable) Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

11. Secondary Outcome: Number of Participants With Favorable Clinical Response in the ME Analysis Set at TOC
Description: The secondary efficacy outcome is favorable clinical response of the patients in the ME (Microbiologically Evaluable) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug.
Population: Patients in CE analysis set with baseline Gram-negative pathogen (= ME (Microbiologically Evaluable) Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

12. Secondary Outcome: Number of Participants With Favorable Clinical Response in the ME Analysis Set at LFU.
Description: The secondary efficacy outcome is favorable clinical response of the patients in the ME (Microbiologically Evaluable) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug
Population: Patients in CE analysis set with baseline Gram-negative pathogen (= ME (Microbiologically Evaluable) Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

13. Secondary Outcome: Number of Participants With Favorable Microbiological Response in the mMITT Analysis Set at EOIV.
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at end of inpatient intravenous therapy (EOIV). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug
Population: Patients in mMITT (Microbiological Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 4 | 2
Participants | 3 | 2

14. Secondary Outcome: Favorable Microbiological Response in the mMITT Analysis Set at TOC.
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug
Population: Patients in mMITT (Microbiological Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 4 | 2
Participants | 3 | 2

15. Secondary Outcome: Number of Participants With Favorable Microbiological Response in the mMITT Analysis Set at LFU.
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug.
Population: Patients in mMITT (Microbiological Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 4 | 2
Participants | 3 | 2

16. Secondary Outcome: Number of Participants With Favorable Microbiological Response in the ME Analysis Set at EOIV.
Description: as for outcome 10
Time Frame: Within 72 hours after administration of the last dose of inpatient IV study drug
Population: Patients in ME (Microbiologically Evaluable) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

17. Secondary Outcome: Number of Participants With Favorable Microbiological Response in the ME Analysis Set at TOC.
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the ME (Microbiologically Evaluable) Analysis Set at test-of-cure (TOC). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 21 to 28 days after the start of inpatient IV study drug
Population: Patients in ME (Microbiologically Evaluable) Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

18. Secondary Outcome: Number of Participants With Favorable Microbiological Response in the ME Analysis Set at LFU
Description: The secondary efficacy outcome is favorable microbiological response of the patients in the ME (Microbiologically Evaluable) Analysis Set at late follow-up (LFU). The clinical outcome has three categories: Favorable clinical response, Clinical failure, and Indeterminate.
Time Frame: 35 to 42 days after the start of inpatient IV study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

19. Secondary Outcome: Number of Participants With Infection-related Mortality in the MITT Analysis Set at TOC
Description: The secondary efficacy outcome is infection-related mortality of the patients in the MITT (Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC).
Time Frame: 21 to 28 days after the start of inpatient IV study drug
Population: Patients in MITT (Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 47 | 50
Participants | 0 | 0

20. Secondary Outcome: Number of Participants With Infection-related Mortality in the MITT Analysis Set at LFU
Description: The secondary efficacy outcome is infection-related mortality of the patients in the MITT (Modified Intent-To-Treat) Analysis Set at late follow-up (LFU).
Time Frame: 35 to 42 days after the start of inpatient IV study drug
Population: Patients in MITT (Modified Intent-to-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 47 | 50
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With Infection-related Mortality the mMITT Analysis Set at TOC
Description: The secondary efficacy outcome is infection-related mortality of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at test-of-cure (TOC).
Time Frame: 21 to 28 days after the start of inpatient IV study drug
Population: Patients in mMITT (Microbiological Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

22. Secondary Outcome: Number of Participants With Infection-related Mortality in the mMITT Analysis Set at LFU.
Description: The secondary efficacy outcome is infection-related mortality of the patients in the mMITT (Microbiological Modified Intent-To-Treat) Analysis Set at late follow-up (LFU).
Time Frame: 35 to 42 days after the start of inpatient IV study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

23. Secondary Outcome: 30 Day All-cause Mortality in the MITT Analysis Set
Description: The secondary efficacy outcome is all-cause mortality of the patients in the MITT (Modified Intent-To-Treat) Analysis Set, which is mortality within 30 days after the last dose of inpatient IV study drug.
Time Frame: 30 days after the last dose of inpatient IV study drug
Population: Patients in MITT (Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 47 | 50
Participants | 2 | 2

24. Secondary Outcome: 30 Day All-cause Mortality in the mMITT Analysis Set
Description: The secondary efficacy outcome is all-cause mortality of the patients in the mMITT (microbiological Modified Intent-To-Treat) Analysis Set, which is mortality within 30 days after the last dose of inpatient IV study drug.
Time Frame: 30 days after the last dose of inpatient IV study drug
Population: Patients in mMITT (Modified Intent-To-Treat) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of the first dose of IV study drug to 30 days following the last dose of study drug. All patients were followed until last follow up which occurred 35-42 days following the first dose of study drug.
Arm/Group | Ceftolozane/Tazobactam Arm | Standard of Care (SOC) Arm
All-Cause Mortality (participants affected / at risk) | 3/47 | 2/50
Serious Adverse Events (participants affected / at risk) | 33/47 | 33/50
Other Adverse Events (participants affected / at risk) | 9/47 | 6/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftolozane/Tazobactam Arm (N=47) | Standard of Care (SOC) Arm (N=50)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 1
Bilirubin increased (Hepatobiliary disorders) | 1 | 0
Bloodstream infection (Infections and infestations) | 5 | 6
Catheter related infection (Infections and infestations) | 4 | 1
Chest pain (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Confusion (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Creatinine increased (Renal and urinary disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 13
Fever (General disorders) | 6 | 8
Headache (Nervous system disorders) | 1 | 1
Heart failure (Cardiac disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Infections and infestations (Infections and infestations) | 3 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Lung infection (Infections and infestations) | 5 | 10
Multi-organ failure (General disorders) | 1 | 1
Papilledema (Eye disorders) | 0 | 1
Pulmonary embolism (Vascular disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Splenic infection (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Viral hepatitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftolozane/Tazobactam Arm (N=47) | Standard of Care (SOC) Arm (N=50)
ALT elevation (Hepatobiliary disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Urinary tract infection (Infections and infestations) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT03485950/Prot_SAP_000.pdf